CLINICAL TRIAL: NCT01112956
Title: Serologic Assays for the Diagnosis of Herpes Simplex Virus Type 2: Development of Testing Strategies
Brief Title: Serologic Assays for the Diagnosis of Herpes Simplex Virus Type 2
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Massachusetts General Hospital (Other); Johns Hopkins University (Other); NYU Langone Health (Other)
Responsible Party: Fujie Xu/Epidemiologist, CDC
Other Study IDs: CDC-NCHHSTP-1127
Record Dates: First submitted 2009-10-13; First posted 2010-04-29 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Genital Herpes
Keywords: HSV-2; HSV-1; Sensitivity; Specificity; Testing algorithm; Test evaluation
MeSH Terms: conditions — Herpes Genitalis; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- STD clinic patients: Patients attending sexually transmitted Disease clinics. If the initial testing result reported to the patient is confirmed by the Western Blot test, no follow-up specimens will be collected. If the initial testing result reported to the patient is different from the result by the Western Blot test, patients will be asked to provide a follow-up specimen 3-4 months after initial testing.
- Pregnant women: Women recruited from prenatal clinic. A follow-up visit may or may not needed depending on results from the initial test and Western blot test.
- Men who have Sex with men (MSM): Men recruited from a clinic for MSM with high risk for HIV infection. A follow-up visit may or may not needed depending on results from the initial test and Western blot test.

SUMMARY:
The purposes of this study are:

* To determine the accuracy of commercially available serologic assays in diagnosing patients with herpes simplex virus type 2 (HSV-2);
* To assess the sensitivity and specificity of the commerical assays using HSV-2 western blot as the "gold standard" in a diverse patient population;
* To develop testing strategies and recommendations for screening asymptomatic populations for HSV-2.

DETAILED DESCRIPTION:
The purposes of this study are:

* To determine the accuracy of commercially available serologic assays in diagnosing patients with herpes simplex virus type 2 (HSV-2);
* To assess the sensitivity and specificity of the commerical assays using HSV-2 western blot as the "gold standard" in a diverse patient population;
* To develop testing strategies and recommendations for screening asymptomatic populations for HSV-2.

We will evaluate the assays in diverse populations:

1. STD clinic population
2. Men who have sex with men, with high prevalence of HIV infection
3. Pregnant women

The study will inform the development of testing strategies:

1. Combine commercial tests to optimize positive predict value (PPV) and negative predict value (NPV)
2. Increase cutoff values to increase PPV
3. Understand factors associated with false positive results that may include HSV-1 infection, pregnancy status, HIV infection, and age/race etc.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 16-55 years of age

Exclusion Criteria:

* Those who refuse to get tested for HIV

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will comprise of diverse ethnic and racial populations derived from 3 Health and Human Services Regions and recruited from different type of clinics: 1) STD clinics 2) Prenatal clinic 3) Health clinic for gay men
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity using Western Blot as the Gold Standard test | Up to 4 months after initial testing

SECONDARY OUTCOMES:
In population with relative low prevalence of HSV-2 infection (e.g. persons <=25 years), whether a combination of tests (i.e. testing algorithm(s)) can increase the positive predictive value to the level of >= 95% | Up to 4 months after initial testing

CONTACTS AND LOCATIONS:
Overall Officials: Donna Felsenstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University School of Medicine, New York, New York